CLINICAL TRIAL: NCT05050318
Title: Collection of Serum Samples From Children 6 Months to < 9 Years of Age Who Received Fluzone® Quadrivalent and Adults ≥ 65 Years of Age Who Received Fluzone® High-Dose Quadrivalent, Influenza Vaccines, 2021-2022 Formulations
Brief Title: Annual Study for Collection of Serum Samples in Children and Older Adults Receiving the 2021-2022 Formulations of Fluzone Quadrivalent Vaccine and Fluzone High-Dose Quadrivalent Vaccine, Respectively
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GRC00102; U1111-1266-5255 (Registry Identifier: ICTRP)
Record Dates: First submitted 2021-09-03; First posted 2021-09-20 (Actual); Results first posted 2022-09-14 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Influenza Immunization; Healthy Volunteers
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Vaccines, Combined

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1: Fluzone Quadrivalent Influenza Vaccine: 6 to <36 Months (Experimental): Participants aged 6 to <36 months received a 0.5-milliliters (mL) dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 1. Participants for whom 2 doses of influenza vaccine were recommended per Advisory Committee on Immunization Practices (ACIP), a second dose was administered at Day 28.
  Interventions: Biological: Fluzone Quadrivalent vaccine, No Preservative (0.5-mL dose), 2021-2022 formulation
- Group 2: Fluzone Quadrivalent Influenza Vaccine: 3 to <9 Years (Experimental): Participants aged 3 to <9 years received a 0.5-mL dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 1. Participants for whom 2 doses of influenza vaccine were recommended per ACIP, a second dose was administered at Day 28.
  Interventions: Biological: Fluzone Quadrivalent vaccine, No Preservative (0.5-mL dose), 2021-2022 formulation
- Group 3: Fluzone High-Dose Quadrivalent Influenza Vaccine: >=65 Years (Experimental): Participants aged >= 65 years received a 0.7-mL dose of Fluzone High-Dose Quadrivalent vaccine intramuscularly at Day 1.
  Interventions: Biological: Fluzone High-Dose Quadrivalent vaccine (0.7-mL dose), 2021-2022 formulation

INTERVENTIONS:
Biological: Fluzone Quadrivalent vaccine, No Preservative (0.5-mL dose), 2021-2022 formulation — Suspension for injection in a pre-filled syringe Route of administration: Intramuscular (IM)
  Other Names: Fluzone® Quadrivalent
  Arms: Group 1: Fluzone Quadrivalent Influenza Vaccine: 6 to <36 Months; Group 2: Fluzone Quadrivalent Influenza Vaccine: 3 to <9 Years
Biological: Fluzone High-Dose Quadrivalent vaccine (0.7-mL dose), 2021-2022 formulation — Suspension for injection in a pre-filled syringe Route of administration: Intramuscular (IM)
  Other Names: Fluzone High-Dose Quadrivalent
  Arms: Group 3: Fluzone High-Dose Quadrivalent Influenza Vaccine: >=65 Years

SUMMARY:
This was a phase IV, multi-center, open-label study. The study collected serum samples from children 6 months to less than (<) 9 years of age who received Fluzone Quadrivalent vaccine and adults greater than or equal to (>=) 65 years of age who received Fluzone High-Dose Quadrivalent vaccine for submission to CBER to aid in the influenza vaccine strain selection process.

DETAILED DESCRIPTION:
Study duration per participant was approximately 28 days for participants with 6 months to < 9 years of age, and 21 days for participants >= 65 years of age, including 1 to 3 visits (1 or 2 vaccination visits) and 1 or 2 telephone calls, depending on study Group.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 months to < 9 years or >= 65 years of age on the day of first study vaccination (study product administration).
* For infants and toddlers, born at full term of pregnancy (>=37 weeks) or born after a gestation period of 27 through 36 weeks.
* For participants 6 to < 12 months of age, born at full term of pregnancy (>= 37 weeks) and with a birth weight >= 5.5 pound (lbs) (2.5 kilogram [kg]).
* Informed consent form (ICF) has been signed and dated by participants >= 65 years of age.
* Assent form has been signed and dated by participants 7 to < 9 years of age, and ICF has been signed and dated by parent(s) or another legally acceptable representative for participants 6 months to < 9 years of age.
* Participants or participant and parent/legally acceptable representative (of participants 6 months to < 9 years of age) were able to attend all scheduled visits and complied with all study procedures.

Exclusion Criteria:

* Participants are excluded from the study if any of the following criteria apply:
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the 3 months preceding planned inclusion).
* Known systemic hypersensitivity to any of the study intervention components, or history of a life-threatening reaction to the study interventions used in the study or to a product containing any of the same substances.
* Thrombocytopenia, contraindicating IM injection, at the discretion of the Investigator.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination.
* Chronic illness that, in the opinion of the Investigator, was at a stage where it might interfere with study conduct or completion.
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of study intervention administration or febrile illness (temperature >= 100.4° Fahrenheit [38.0° Celsius]). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Alcohol, prescription drug, or substance abuse that, in the opinion of the Investigator, might interfere with the study conduct or completion.
* History of serious adverse reaction to any influenza vaccine.
* Personal history of Guillain-Barré syndrome.
* Any condition that in the opinion of the Investigator would pose a health risk to the participant if enrolled or could interfere with the evaluation of the vaccine.
* Personal history of clinically significant developmental delay (at the discretion of the Investigator), neurologic disorder, or seizure disorder.
* Known seropositivity for human immunodeficiency virus, hepatitis B, or hepatitis C.
* Receipt of any vaccine in the 30 days preceding the first study intervention administration, or planned receipt of any vaccine before Visit 2 for participants receiving 1 dose of influenza vaccine or Visit 3 for participants receiving 2 doses of influenza vaccine.
* Previous vaccination against influenza (in the 2021-2022 influenza season) with an investigational or marketed vaccine.
* Receipt of blood-derived immune globulins, blood, or blood-derived products in the past 3 months.
* Participation at the time of study enrollment (or in the 30 days preceding the first study vaccination) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure.

Note: Participants might be considered eligible for enrollment if no intervention for the other study occurred within the 30 days prior to the first study vaccination and none were planned before the participant would complete safety surveillance for the present study.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (2):
- United States (2):
  - Investigational Site Number :8400001, Bardstown, Kentucky
  - Investigational Site Number :8400002, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: GRC00102 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25271&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 08 September 2021 to 20 September 2021 at 2 active sites in the United States.
Pre-assignment Details: A total of 90 participants were enrolled in the study.
Groups:
- Group 1: Fluzone Quadrivalent Influenza Vaccine: 6 to <36 Months: Participants aged 6 to less than (<) 36 months received a 0.5-milliliters (mL) dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 1. Participants for whom 2 doses of influenza vaccine were recommended per Advisory Committee on Immunization Practices (ACIP), a second dose was administered at Day 28.
- Group 3: Fluzone High-Dose Quadrivalent Influenza Vaccine: >=65 Years: Participants aged greater than or equal to (>=) 65 years received a 0.7-mL dose of Fluzone High-Dose Quadrivalent vaccine intramuscularly at Day 1.
Period: Overall Study
Arm/Group | Group 1: Fluzone Quadrivalent Influenza Vaccine: 6 to <36 Months | Group 2: Fluzone Quadrivalent Influenza Vaccine: 3 to <9 Years | Group 3: Fluzone High-Dose Quadrivalent Influenza Vaccine: >=65 Years
Started | 29 | 31 | 30
Vaccinated | 28 | 31 | 30
Completed | 28 | 31 | 30
Not Completed | 1 | 0 | 0
Not completed — Protocol Deviation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all vaccinated participants which included all participants who had received at least 1 dose of the study vaccine.
Groups:
- Group 1: Fluzone Quadrivalent Influenza Vaccine: 6 to <36 Months: Participants aged 6 to <36 months received a 0.5-mL dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 1. Participants for whom 2 doses of influenza vaccine were recommended per ACIP, a second dose was administered at Day 28.
- Total: Total of all reporting groups
Arm/Group | Group 1: Fluzone Quadrivalent Influenza Vaccine: 6 to <36 Months | Group 2: Fluzone Quadrivalent Influenza Vaccine: 3 to <9 Years | Group 3: Fluzone High-Dose Quadrivalent Influenza Vaccine: >=65 Years | Total
Number analyzed (Participants) | 28 | 31 | 30 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28 | 31 | 0 | 59
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 30 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.83 (0.410) | 4.81 (1.83) | 73.3 (4.31) | 27.0 (33.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 15 | 40
  Male | 17 | 17 | 15 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 0 | 4
  White | 26 | 28 | 30 | 84
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Aged 6 Months to <9 Years Who Provided Serum Samples for Analysis: Groups 1 and 2
Description: Blood samples were collected from participants at first vaccination at Visit 1 (Day 1; pre-vaccination) and at Day 28 after final vaccination either at Visit 2 (Visit 1 + 28 days) for participants who received 1 dose of influenza vaccine; or at Visit 3 (Visit 2 + 28 days) for participants who received 2 doses of influenza vaccine as recommended by ACIP. Collected blood samples were provided to Center for Biologics Evaluation and Research (CBER) for further analysis by World Health Organization (WHO), Centers for Disease Control and Prevention (CDC), and Food and Drug Administration (FDA) to support formulation recommendations for subsequent influenza vaccines.
Time Frame: Visit 1 (Day 1; pre-vaccination) and 28 days post-final vaccination at Visit 2 (for participants with 1 vaccination)/Visit 3 (for participants with 2 vaccination)
Population: Analysis was performed on all vaccinated participants. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Fluzone Quadrivalent Influenza Vaccine: 6 to <36 Months | Group 2: Fluzone Quadrivalent Influenza Vaccine: 3 to <9 Years
Number analyzed (Participants) | 28 | 31
Participants
  Visit 1 | 28 | 31
  Visit 2: number analyzed (Participants) | 20 | 31
  Visit 2 | 20 | 31
  Visit 3: number analyzed (Participants) | 7 | 0
  Visit 3 | 7 | 0

2. Primary Outcome: Number of Participants Aged >=65 Years Who Provided Serum Samples for Analysis: Group 3
Description: Blood samples were collected from participants at first vaccination at Visit 1 (Day 1; pre-vaccination) and 21 days after vaccination (Visit 2). Collected blood samples were provided to CBER for further analysis by WHO, CDC, and FDA to support formulation recommendations for subsequent influenza vaccines.
Time Frame: Visit 1 (Day 1; pre-vaccination) and 21 days post-vaccination (Visit 2)
Population: Analysis was performed on all vaccinated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 3: Fluzone High-Dose Quadrivalent Influenza Vaccine: >=65 Years
Number analyzed (Participants) | 30
Participants
  Visit 1 | 30
  Visit 2 | 30

ADVERSE EVENTS:
Time Frame: Reported adverse events (AE) data were collected from Visit 1 (Day 1) up to end of the study (i.e., up to Day 21 for adult participants [>=65 years], up to Day 28 for child participants [6 to <9 years] who received 1 dose and up to Day 56 for participants who received 2 doses).
Description: Analysis was performed on all vaccinated participants.
Groups:
- Group 3: Fluzone High-Dose Quadrivalent Influenza Vaccine: >=65 Years: Participants aged >=65 years received a 0.7-mL dose of Fluzone High-Dose Quadrivalent vaccine intramuscularly at Day 1.
Arm/Group | Group 1: Fluzone Quadrivalent Influenza Vaccine: 6 to <36 Months | Group 2: Fluzone Quadrivalent Influenza Vaccine: 3 to <9 Years | Group 3: Fluzone High-Dose Quadrivalent Influenza Vaccine: >=65 Years
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 0/28 | 0/31 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT05050318/Prot_SAP_000.pdf